CLINICAL TRIAL: NCT01526525
Title: Effect of Perioperative Electroacupuncture With Tramadol and Ketamine on Postoperative Analgesia in Prostatectomy: a Randomized Placebo-controlled Trial
Brief Title: Perioperative Electroacupuncture on Postoperative Analgesia in Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, NTRITSOU VAGIA, MD, ANESTHESIOLOGIST, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6151/ 22-7-2009
Record Dates: First submitted 2012-01-28; First posted 2012-02-06 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Pain, Postoperative
Keywords: tramadol; ketamine; parecoxib; paracetamol; numerical rating scale (NRS); McGill (SF-MPQ); electronic pressure algometer; Spielberger State Trait Anxiety Inventory STAI Y-6 item
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Ketamine; Morphine; parecoxib; Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TK (Placebo Comparator): In TK group when the closure of the abdominal walls started, a certified acupuncturist expert put needles, Ener-Qi 0.26Χ25mms, in LI4 point in both hands, the needles were not inserted in the skin but they were put atop the skin and were secured by adhesive tape. For 30min in the E/A stimulator ITO ES-160 the indicator light was on but no electrical current was applied. Thereafter the E/A device deactivated and after the awakening of the patients, it was connected in ST36 and LI4 points for 30min with the same technique. The electrodes were connected to each other in every point, as the right with the left point of LI4 and the right with the left point of ST36. The patients were told that they may or may not feel electrical current because of its very high frequency.
  Interventions: Drug: Tramadol; Drug: Ketamine; Drug: Morphine; Procedure: sedation; Procedure: rescue analgesia; Drug: Parecoxib; Drug: paracetamol
- TKE (Active Comparator): In TKE group when the closure of the abdominal walls started, a certified acupuncturist expert put needles, Ener-Qi 0.26Χ25mms, in LI4 point at 2cm depth in both hands and E/A was applied for 30min with the E/A stimulator ITO ES-160 in constant pulse program with 300μs duration and 100Hz frequency. After the needles were connected to the E/A stimulator, they were secured by adhesive tape. The response which certified the right needle placement was the adjacent muscular twitch. Thereafter the E/A device was deactivated and after the awakening of the patients, E/A was administered in ST36 and LI4 points for 30min with 4Hz frequency. The electrodes were connected to each other in every point, as the right with the left point of LI4 and the right with the left point of ST36.
  Interventions: Drug: Tramadol; Drug: Ketamine; Drug: Morphine; Procedure: sedation; Procedure: rescue analgesia; Drug: Parecoxib; Drug: paracetamol

INTERVENTIONS:
Drug: Tramadol — Tramadol 1.5mg/kg bolus IV 30min before the end of the surgery and co instantaneously the CIV infusion of tramadol 0.15mg/kg/h started with continuous infusion in an adjustable flow disposable pump (paragon®)
Drug: Ketamine — ketamine 10mg bolus IV 30min before the end of the surgery and co instantaneously the CIV infusion of ketamine, in subanesthetic doses, 0,15mg/kg/h started with continuous infusion in an adjustable flow disposable pump (paragon®). Ketamine's dose was altered so as not to exceed the 300mg/24h.
Drug: Tramadol — If NRS scale was ≥3, PPI scale ≥2 and the algometer count ≤0,5Kg it was assumed as a non acceptable pain treatment. Tramadol 50mg IV bolus was firstly administered to the patients.The aim was that the Tramadol 24h dose would not exceed 600mg
Drug: Morphine — If NRS scale was ≥3, PPI scale ≥2 and the algometer count ≤0,5Kg it was assumed as a non acceptable pain treatment. Tramadol 50mg IV bolus was firstly administered to the patients and if the NRS scale was not decreased at least about 2 points after 30 minutes, morphine 2mg IV was then administered and it could be repeated
Procedure: sedation — If the patient had sedation score >2 then the analgesic infusion would be stopped, the patient would be assessed again in 1 hour and the infusion would start with the same or decreased flow.
Procedure: rescue analgesia — Meanwhile - 45min,2h,6h,12h and 24h- if the patients had acute pain, the physician would call the anesthesiologist and a new assessment would take place with the relative interventions.
Drug: Parecoxib — An hour before the end of the surgery all patients were administered with parecoxib 40mg (IV)
Drug: paracetamol — 30min before the end of the surgery paracetamol 20mg/kg (IV).

SUMMARY:
The aim of the present study is the comparison of the efficacy of the perioperative application of a multimodal analgesia model to the patients, combing common used analgesics via intravenous (IV) route, such as tramadol and ketamine, with or without the Electroacupuncture (E/A) technique application and the frequency of side effects accession.

DETAILED DESCRIPTION:
Seventy patients were scheduled for radical prostatectomy, were recruited to this prospective single-blind, were randomized and placebo-controlled by trial. They were randomly divided into two groups of 35 patients each by a computer-generated randomization sequence, the TKE (Tramadol + Ketamine + Electroacupuncture), and TK (Tramadol + Ketamine + placebo Electroacupuncture.The randomization performed by the certified acupuncturist.

Patients were anesthetized with the same protocol by five anesthesiologists, who were not involved in the postoperative assessment of the patients, but were aware in which group acupuncture was used and in which not. Both groups, TKE and TK, were administered tramadol 1.5mg/kg and ketamine 10mg bolus IV 30min before the end of the surgery and co instantaneously the CIV infusion of tramadol 0.15mg/kg/h and ketamine, in subanesthetic doses, 0.15mg/kg/h started with continuous infusion in an adjustable flow disposable pump (paragon®).Ketamine's dose was altered so as not to exceed the 300mg/24h. An hour before the end of the surgery all patients were administered with parecoxib 40mg (IV) and 30min before paracetamol 20mg/kg (IV).

In TKE group when the closure of the abdominal walls started, a certified acupuncturist expert put needles, Ener-Qi 0.26Χ25mms, in LI4 point at 2cm depth in both hands and E/A was applied for 30min with the E/A stimulator ITO ES-160 in constant pulse program with 300μs duration and 100Hz frequency. After the needles were connected to the E/A stimulator, they were secured by adhesive tape. The response which certified the right needle placement was the adjacent muscular twitch. Thereafter the electroacupuncture machine was deactivated and after the awakening of the patients, E/A was administered in ST36 and LI4 points for 30min with 4Hz frequency. The electrodes were connected to each other in every point, as the right with the left point of LI4 and the right with the left point of ST36. In the TK group the needles were not inserted in the skin but they were put atop the skin and were secured by adhesive tape, the indicator light was on but no electrical current was applied. The patients were told that they may or may not feel electrical current because of its very high frequency.

The study was single blind as patients although they were informed for the Electroacupuncture (E/A) technique during the first session they were anesthetized and the second one was after the awakening of anesthesia and they didn't understand it. On the other hand anaesthesiologists and the certified acupuncturist during the EAc application knew in which group patients belong although they did not deal with them postoperatively. However, patient assessments were performed at standard time points as 45 min in recovery and at 2 h, 6 h, 12 h and 24 h after surgery in the ward by another anaesthesiologist who was not present during the surgery or the recovery room for the first 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Male patient is over 18 years old, especially 50-75 years old
* Patient scheduled for a non-emergency operation
* Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion Criteria:

* Patient receiving monoamine oxidase inhibitors and selective serotonin reuptake inhibitors
* Patient with significant cardiovascular, pulmonary, renal or hepatic disease
* Patient with epilepsy non controlled with treatment or history of seizures
* Patient with morbid obesity (BMI>35)
* Patient with history of chronic opioid exposure
* Patient with history of chronic pain
* Patient with history of postoperative nausea and vomiting
* Patient with cognitive dysfunction
* Patient with history of previous usage of the acupuncture technique
* Patient Greek speaking
* Patient is participating in another clinical trial which may affect this study's outcomes
* Patient with metastatic cancer

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
PAIN SCALES | 45min, 2h, 6h, 12h and 24h following the surgery
  Numerical Rating Scale (NRS) 0-10,from 0=no pain to 10=worst pain imaginable. Present Pain Intensity (PPI) 0-5,from 0= no pain to 5= excruciating. McGill pain scale (SF-MPQ) 0-3,from 0=no pain to 3=severe pain
PATIENTS PAIN THRESHOLD WITH ELECTRONIC PRESSURE ALGOMETER | 45min, 2h, 6h, 12h and 24h following the surgery
  The electronic pressure algometer device was applied 2cm bilateral the middle of the midline extraperitoneal lower abdominal incision and were recorded the pain threshold. It converted in Kg
NUMBER OF PARTICIPANTS WITH ADVERSE EVENTS | 45min, 2h, 6h, 12h and 24h following the surgery
  Nausea:yes/no vomiting:yes/no pruritus:yes/no bowel movement:yes/no Sedation scale 0-3, from 0= awake or sleepy that answers to the questions to 3=asleep who doesn't awake not even with a prod
PATIENTS RESCUE ANALGESIA | 45min, 2h, 6h,12h and 24h following the surgery
  If NRS scale was ≥3, PPI scale ≥2 and the algometer count ≤0,5Kg it was assumed as a non acceptable pain treatment. Tramadol 50mg IV bolus was firstly administered to the patients and if the NRS scale was not decreased at least about 2 points after 30 minutes, morphine 2mg IV was then administered and it could be repeated. The aim was that the Tramadol 24h dose would not exceed 600mg. So with rescue analgesia, tramadol or morphine in mg, we count the total amount of opioids administered
CORTIZOL | : 1st at 8am at the day of the surgery (Cort1), 2nd 45min after the end of the surgery (Cort2) and 3rd at 8am the first postoperative day (Cort3)
  Cortizol levels: ug/dl

SECONDARY OUTCOMES:
PATIENTS WELLBEING, | Preoperatively and 24h following the surgery
  Spielberger State Trait Anxiety Inventory (STAI Y-6 item) 1-4, where 1=not at all and 4 =very much so.
SATISFACTION | 24h following the surgery
  Verbal Rating Scale (VRS) with 6 levels of satisfaction 1-6,from 1=very dissatisfied to 6= very satisfied
SLEEP DISORDERS | 24h following the surgery
  Answer to questions such as "if they slept well?" yes/no "they had nightmares or bad dreams?" yes/no

CONTACTS AND LOCATIONS:
Overall Officials: VAGIA NTRITSOU, Principal Investigator — G.Gennimatas General Hospital; DIMITRIOS VASILAKOS, Study Director — Aristotle University Of Thessaloniki; GEORGIOS DIMITRIADIS, Study Director — G.Gennimatas General Hospital; CHRISTOS KOSTOGLOU, MD, Principal Investigator — G.Gennimatas General Hospital
Locations (1):
- G.Gennimatas GENERAL HOSPITAL OF THESSALONIKI, Thessaloniki, Greece

REFERENCES:
- [Derived] Ntritsou V, Mavrommatis C, Kostoglou C, Dimitriadis G, Tziris N, Zagka P, Vasilakos D. Effect of perioperative electroacupuncture as an adjunctive therapy on postoperative analgesia with tramadol and ketamine in prostatectomy: a randomised sham-controlled single-blind trial. Acupunct Med. 2014 Jun;32(3):215-22. doi: 10.1136/acupmed-2013-010498. Epub 2014 Jan 30. PMID 24480836